CLINICAL TRIAL: NCT03968159
Title: Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Adjunctive Pimavanserin in Subjects With Major Depressive Disorder and Inadequate Response to Antidepressant Treatment (ACP-103-054/059)
Brief Title: Adjunctive Pimavanserin in Subjects With Major Depressive Disorder and Inadequate Response to Antidepressant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-054/059; 2018-003251-37 (EudraCT Number); NCT03999918 (obsolete NCT alias)
Record Dates: First submitted 2019-05-13; First posted 2019-05-30 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Adjunctive Treatment of Major Depressive Disorder
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug - pimavanserin (Experimental): Pimavanserin 34 mg tablets
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg (provided as 2×17 mg tablets) administered orally as a single dose once daily
  Arms: Drug - pimavanserin
Drug: Placebo — Placebo (2×placebo tablets [size- and color-matched to pimavanserin]) administered orally as a single dose once daily
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of adjunctive pimavanserin compared to placebo in subjects with major depressive disorder who have an inadequate response to antidepressant therapy

DETAILED DESCRIPTION:
Two separate studies, idential in design, were planned and initiated under 2 protocol IDs and NCTs, i.e. study ACP-103-54 (NCT03999918) and ACP-103-059 (NCT03968159). In March 2020, recruitment of new patients was paused due to the emerging coronavirus disease 2019 (COVID-19) pandemic. At that point in time, about half of the planned patients had been randomized. The Sponsor decided to combine the 2 identically designed trials, with a prespecified combined statistical analysis plan. As a result, both trials were closed and proceeded with database lock and statistical analysis of the combined data. No further patients were enrolled.

This entry now includes the combined data of studies ACP-103-054 and ACP-103-059.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged 18 years and above
2. A clinical diagnosis of major depressive disorder (MDD)
3. Is being treated with one of the following SSRI or SNRI antidepressants:

   1. Citalopram
   2. Escitalopram
   3. Paroxetine
   4. Fluoxetine
   5. Sertraline
   6. Duloxetine
   7. Venlafaxine
   8. Desvenlafaxine
   9. Venlafaxine XR
4. Inadequate response to SSRI/SNRI antidepressant treatment is confirmed
5. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential OR must agree to use acceptable methods of contraception

Exclusion Criteria:

1. Has a history of psychotic disorder or is currently being treated or requires treatment for post-traumatic stress disorder, acute stress disorder, panic disorder, or obsessive compulsive disorder
2. Has current evidence of delirium or an unstable neurological, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies that would affect the patient's ability to participate in the program
3. Has a known history or symptoms of long QT syndrome
4. Is determined to be inappropriate for the study for any reason

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (41):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - CNS Network, Garden Grove, California
  - Behavioral Research Specialists, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Irvine Clinical Research, Irvine, California
  - Synergy San Diego, Lemon Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Clinical Neuroscience Solutions ( CNS Healthcare)-Jacksonville, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Florida Research Center, Inc., Miami, Florida
  - CNS Health Care (Orlando), Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Synexus Clinical Research, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Collective Medical Research, LLC, Prairie Village, Kansas
  - Clinical Trials of America (Monroe, LA), Monroe, Louisiana
  - Adams Clinical, Watertown, Massachusetts
  - St. Charles Psychiatric Associates-Midwest Research Group, Saint Charles, Missouri
  - Integrative Clinical Trials, Brooklyn, New York
  - Social Psychiatry Research Institute (SPRI), Brooklyn, New York
  - Mount Sinai Hospital, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lake Clinical Research, Rochester, New York
  - Clinical Trial of America, LLC, Hickory, North Carolina
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Clinical Neuroscience Solutions CNS Healthcare, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Future Search Trials of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - IPC Research, Waukesha, Wisconsin
- Finland (5):
  - ARTES Psykiatrinen Palvelukeskus Oy (Mederon Ltd.), Helsinki
  - Savon Psykiatripalvelu Oy, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu Oy at Mehiläinen Pori, Pori
  - Psykiatri- ja psykologikeskus Mentoria, Tampere
- Poland (6):
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski, Bełchatów
  - Przychodnia Śródmieście Sp. z o.o., Bydgoszcz
  - Indywidualna Specijalistyczna Praktyka Lekarska Wiesław Jerzy Cubała, Gdansk
  - Nzop Mentis, Leszno
  - Neurologiczny NZOZ im. dr n. med. Hanki, Plewiska
  - Zachodniopomorski Instytut Psychoterapii, Szczecin
- Russia (8):
  - Mental Health Research Center, Department #6, Moscow
  - St. Nicholas the Wonder Worker Psychiatric Hospital, Saint Petersburg
  - Psychoneurological Dispensary # 5, Saint Petersburg
  - City Narcology Hospital, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Saratov City Clinical Hospital # 2 n.a. V.I. Razumovsky, Saratov
  - Regional Clinical Psychiatric Hospital of St. Sofia, Saratov
  - LION-MED, Voronezh
- Serbia (7):
  - Clinical Center of Serbia, Clinic for psychiatry, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic, Belgrade
  - Special hospital for psychiatric diseases "Kovin", Kovin
  - Clinical Center Kragujevac , Clinic for Psychiatry, Kragujevac
  - Clinical Center Kragujevac, Kragujevac
  - Centre for Mental Health Protection, Clinical Center Nis, Niš
  - Clinical Centre Nis, Clinic for Psychiatry Gornja, Toponica
- Slovakia (3):
  - EPAMED s r.o., Košice
  - Liptovska nemocnice s poliklinikou MUDr. Ivana Stodolu, Psychiatricke oddelenie, Liptovský Mikuláš
  - Centrum Zdravia R.B.K., s.r.o., Svidník
- South Africa (4):
  - Cape Trial Centre, Cape Town
  - Dr DG Dennis Incorporated Knighton Surgery, Cape Town
  - Flexivest Fourteen Research Centre, Unit 1, Durbanville Health Center, Durbanville
  - Dr GP Bosch Clinical Research, Pretoria
- Ukraine (8):
  - Regional Centre of Psychosomatic Disorders based on Psychoneurology Department, Communal Institution "Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnykov, Dnipro
  - Institute of neurology, Psychiatry and Narcology of NAMS of Ukraine, MC "Neuron", Kharkiv
  - Kyiv Railway Clinical Hospital № 1 of Branch "Health Center" of the Public joint stock company "Ukrainian Railway", Kyiv
  - Odesa Regional Medical Centre of Mental Health, Odesa
  - Kherson Regional Psychiatric Hospital Department # 3 and # 10 Kherson region, Stepanovka
  - Ternopil Regional Communal Clinical Psychoneurological Hospital, psychiatric department # 2 (men), psychiatric department # 6 (women), Ternopil State Medical University n.a. I.Y. Gorbachevskyy, Chair of Psychiatry, Narcology and Medical Psychology, Ternopil
  - Communal Institution "Vinnytsia Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Department #7 (male), Department #10 (female),Vinnytsia National Medical University n.a. M.I.Pyrogov, Department of Psychiatry, Narcology and Psychotherapeuti, Vinnytsia
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Male Department #14, Female Department #15, Vinnytsya National Medical University n.a. M.I.Pyrogov, Department of Psychiatry, Narcology and Psychotherapeutic, Vinnytsia
- United Kingdom (3):
  - MAC Clinical Research - Blackpool, Blackpool
  - MAC Clinical Research Ltd - Liverpool, Liverpool
  - MAC Clinical Research - Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in patients with with major depressive disorder who had an inadequate response to antidepressant treatment.
Pre-assignment Details: During the screening period, patients were assessed for study eligibility, and prohibited medications were discontinued when medically appropriate.
Groups:
- Pimavanserin: Pimavanserin 34 mg administered orally as a single dose once daily
- Placebo: Placebo tablets administered orally as a single dose once daily
Period: Overall Study
Arm/Group | Pimavanserin | Placebo
Started | 148 | 150
Completed | 135 | 135
Not Completed | 13 | 15
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Use of prohibited medication | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Not further specified | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimavanserin | Placebo | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.45) | 44.5 (14.92) | 45.8 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 112 | 208
  Male | 52 | 38 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 137 | 137 | 274
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148
  Finland | 3 | 9 | 12
  Poland | 12 | 6 | 18
  Russia | 18 | 12 | 30
  Serbia | 9 | 8 | 17
  Slovakia | 4 | 3 | 7
  South Africa | 1 | 1 | 2
  Ukraine | 14 | 16 | 30
  United Kingdom | 13 | 21 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 5 in Hamilton Depression Scale (17 Items) (HAMD-17) Total Score
Description: The HAMD-17 consists of 8 items with a score on a 3 point scale and 9 items with a score on a 5 point scale. The total score ranging from 0 to 52 will be calculated as the sum of the scores for all 17 items. Higher total scores denote more severe depression.
Time Frame: Baseline, Week 5
Population: Full Analysis Set: all subjects who were randomized, received at least one dose of study drug, and had a baseline value and at least one postbaseline value for HAMD-17 total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -9.0 (0.58) | -8.1 (0.58)
Statistical Analysis 1: Comparison: Pimavanserin vs Placebo; Test type: Superiority; p = 0.2956, Mixed-effects model for repeated measure; LSM difference = -0.9, 95% CI 2-sided [-2.5 to 0.8], Standard Error of Mean 0.82

2. Secondary Outcome: Change From Baseline to Week 5 in Clinical Global Impression-Severity (CGI-S) Score for Depressive Symptoms
Description: The CGI-S rates the severity of a subject's depression over the past 7 days and the score ranges from 1 to 7. Higher CGI-S scores denote more severe depression.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -1.4 (0.10) | -1.1 (0.10)

3. Secondary Outcome: Change From Baseline to Week 5 in Sheehan Disability Scale (SDS) Score
Description: The SDS is a 3-item subject-facing questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. Subjects rate each item using an 11-point scale ranging from 0 (not at all) to 10 (extremely). Higher scores denote greater disability.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -2.5 (0.22) | -2.1 (0.22)

4. Secondary Outcome: Change From Baseline to Week 5 in the Changes in Sexual Functioning Questionnaire Short Form
Description: The CSFQ-14 is a 14-item version of the CSFQ. This is a patient-facing questionnaire, with a male version and a female version. The total score ranging from 14 to 70 will be calculated as the sum of the scores for all 14 items. Higher total scores denote better sexual functioning.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | 3.4 (0.66) | 2.5 (0.66)

5. Secondary Outcome: Change From Baseline to Week 5 in Karolinska Sleepiness Scale (KSS) Score
Description: The KSS is a scale that measures the subject's drowsiness and is frequently used in studies measuring subjective sleepiness. Scoring is based on a 9-point verbally anchored scale going from "1 = extremely alert" to "9 = very sleepy, great effort to keep awake, fighting sleep". Higher scores denote more drowsiness.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -1.4 (0.15) | -0.8 (0.15)

6. Secondary Outcome: Change From Baseline to Week 1 in the HAMD-17 Total Score
Description: as for outcome 1
Time Frame: Baseline, 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -3.8 (0.34) | -3.2 (0.34)

7. Secondary Outcome: Treatment Responder and Treatment Remission Rates at Week 5
Description: The HAMD-17 consists of 8 items with a score on a 3 point scale and 9 items with a score on a 5 point scale. The total score ranging from 0 to 52 will be calculated as the sum of the scores for all 17 items. Treatment response is defined as a reduction from Baseline in HAMD-17 total score of 50% or more. Treatment remission is defined as a HAMD-17 total score ≤7.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
Participants
  Responder | 46 | 46
  Remitter | 27 | 25

8. Secondary Outcome: Change From Baseline to Week 5 in the Hamilton Depression (HAMD) Anxiety/Somatization Factor Score
Description: The Anxiety/Somatization factor of the HAMD-17 includes 6 items: psychic anxiety, somatic anxiety, gastrointestinal somatic symptoms, general somatic symptoms, hypochondriasis, and insight. The HAMD-17 Anxiety/Somatization factor score ranging from 0 to 18 will be calculated as the sum of the scores for the 6 items. Higher scores denote more severe anxiety/somatization condition.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -2.5 (0.21) | -2.5 (0.21)

9. Secondary Outcome: Change From Baseline to Week 5 in the Barratt Impulsiveness Scale (BIS-11)
Description: The BIS-11 is a questionnaire designed to assess the personality/behavioral construct of impulsiveness. It is composed of 30 items describing common impulsive or non-impulsive (reverse scored items: 1, 7, 8, 9, 10, 12, 13, 15, 20, 29, and 30) behaviors and preferences. Items are scored on the following 4-point scale: Rarely/Never = 1; Occasionally = 2; Often = 3; Almost Always/Always = 4. For reverse scored items, a response of 1 is recoded to 4; 2 is recoded to 3; 3 is recoded to 2; and 4 is recoded to 1. The BIS-11 score ranging from 30 to 120 will be calculated as the sum of the scores for all 30 items. Higher scores denote more impulsiveness.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | -3.0 (0.64) | -2.5 (0.64)

10. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score for Depressive Symptoms at Week 5
Description: The CGI-I rates the change in a subject's depression over the past 7 days relative to the subject's symptoms at Baseline and the score ranges from 1 to 7. Higher CGI-I scores denote less improvement in Depression.
Time Frame: Baseline, 5 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 148 | 149
score on a scale | 2.7 (0.09) | 2.9 (0.09)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were to be documented through 30 days after the last planned dose in the study which was to be administered at Week 6.
Arm/Group | Pimavanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/150
Serious Adverse Events (participants affected / at risk) | 2/148 | 2/150
Other Adverse Events (participants affected / at risk) | 54/148 | 43/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=148) | Placebo (N=150)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=148) | Placebo (N=150)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 9 (9)
Headache (Nervous system disorders) | 31 (49) | 27 (39)

LIMITATIONS AND CAVEATS:
In March 2020, recruitment of new patients was paused due to the emerging coronavirus disease 2019 (COVID-19) pandemic. At that point in time, about half of the planned patients had been randomized. The Sponsor decided to combine this trial with the identically designed trial ACP-103-054, with a prespecified combined statistical analysis plan. As a result, both trials were closed and proceeded with database lock and statistical analysis of the combined data. No further patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's Prior written consent. At least 60 days prior to submitting a manuscript or Prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (3):
  • Study Protocol: Study ACP-103-059 protocol (NCT03968159) (2020-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03968159/Prot_000.pdf
  • Study Protocol: Study ACP-103-054 protocol (NCT03999918) (2020-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03968159/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03968159/SAP_001.pdf